CLINICAL TRIAL: NCT02498158
Title: Functional Neural Connectivity at Rest, as a Diagnostic Tool for Intolerance to Heat and Return to Duty After Exertional Heat Stroke
Brief Title: Functional Neural Connectivity at Rest as a Diagnostic Tool for Intolerance to Heat
Acronym: fMRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2380-15-SMC
Record Dates: First submitted 2015-07-12; First posted 2015-07-15 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Functional Neural Connectivity
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- experimental protocol: Functional neural connectivity at rest of 3 groups (heat tolerant, heat intolerant and healthy subjects) will be assessed using the anatomical and functional MRI scans and compared.
  Interventions: Device: MRI scans

INTERVENTIONS:
Device: MRI scans — 20 subject (10 tolerant and 10 intolerant to heat) will undergo MRI scans (GE healthcare manufacturer) as follows:
  1. anatomical scan according to standard protocol
  2. functional scan according to the standard protocol of rest-state fMRI.
  scans of 10 healthy subjects will be taken from existing scans at the imaging department.

SUMMARY:
Functional neural connectivity at rest of 3 groups (heat tolerant, heat intolerant and healthy subjects) will be assessed using the anatomical and functional MRI scans and compared.

DETAILED DESCRIPTION:
20 healthy subjects that had already underwent Heat Tolerance Test (HTT) at the Heller Institute of Medical Research (Sheba Medical Center) will be recruited and divided into 2 groups: heat tolerant and heat intolerant (according to the HTT results). They will be asked to arrive to one experimental day at the imaging department in Sheba Medical Center and undergo anatomical and functional MRI scans.

Third group will consist of 10 existing brain scans (separated from personal details) of healthy males, at the same age range and who had never gone through heat injury.

Data will be analysed by fMRI expert in order to compare the functional neural connectivity at rest between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy subjects
* underwent heat injury in the past two months
* underwent Heat Tolerance Test at the Heller Institute of Medical research

Exclusion Criteria:

* drug or alcohol use
* history of neurological disorders, mental retardation or head injury
* history or diagnosis of psychiatric disorders
* claustrophobia

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: population of soldiers from the israeli defence forces (IDF), healthy in general, who had gone through heat injury (heat fatigue or hyperthermia) in the two month prior to their recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
functional neural connectivity | one day
  MRI scans will be interpreted by fMRI expert and then compared between heat tolerant and intolerant subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Frenkel, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel